CLINICAL TRIAL: NCT04852900
Title: Effects of Different Dosage of Decompression Therapy on Symptoms of Lumbar Radiculopathy
Brief Title: Different Dosage of Decompression Therapy on Symptoms of Lumbar Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/00856 Iqra Hamid
Record Dates: First submitted 2021-04-20; First posted 2021-04-21 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Lumbar Radiculopathy
Keywords: Pain; Radiculopathy; Lumbar; Decompression
MeSH Terms: conditions — Radiculopathy; Pain | interventions — Decompression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Decompression with 30% (Experimental): Decompression with 30% and mobilization
  Interventions: Other: Decompression with 30%
- Decompression with 40% (Experimental): Decompression with 40% and mobilization
  Interventions: Other: Decompression with 40%
- Decompression with 50% (Experimental): Decompression with 50% and mobilization
  Interventions: Other: Decompression with 50%

INTERVENTIONS:
Other: Decompression with 30% — * Hot Pack for 10 mins Soft Tissue Mobilization
  * Muscle Strengthening
  * Decompression with 30% The total time for the session will be 45 minutes and there will be 03 sessions/week for 6 weeks
  Arms: Decompression with 30%
Other: Decompression with 40% — * Hot Pack for 10 mins Soft Tissue Mobilization
  * Muscle Strengthening
  * Decompression with 30% The total time for the session will be 45 minutes and there will be 03 sessions/week for 6 weeks
  Arms: Decompression with 40%
Other: Decompression with 50% — * Hot Pack for 10 mins Soft Tissue Mobilization
  * Muscle Strengthening
  * Decompression with 30% The total time for the session will be 45 minutes and there will be 03 sessions/week for 6 weeks
  Arms: Decompression with 50%

SUMMARY:
This study will provide evidence about how much dose of decompression more effective for the treatment of lumbar radiculopathy. As this hypothesis has no evidence about the dosage of decompression in literature till now.

DETAILED DESCRIPTION:
Decompression therapy differs from traction-based therapy in that the traction applied to the spine in decompression therapy is typically alternated between lower and higher levels of tension for predetermined periods of time. In either therapy, spinal tension is maintained for the period's typically extending 30-minutes or longer. This study will provide evidence about how much dose of decompression more effective for the treatment of lumbar radiculopathy. As this hypothesis has no evidence about the dosage of decompression in literature till now.

ELIGIBILITY:
Inclusion Criteria:

* Both Genders
* Age between 30 to 50 years
* Unilateral Radiculopathy
* Limited SLR (Less than 60 degree)
* Pain on Numeric Pain Rating Scale < 7
* BMI ≤ 30

Exclusion Criteria:

* Severe paraspinal Muscle Spasm
* Acute prolapse intervertebral disc
* Bilateral Positive SLR
* Osteoporotic
* H/O Spinal Fracture

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-07-10 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 6th week
  The Numeric Pain Rating Scale (NPRS) (an outcome measure) that is a uni-dimensional measure of pain intensity in adults(21). The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
SLR through Inclinometer | 6th week
  The Straight Leg Raise (SLR) test is a neurodynamic test. Neurodynamic tests check the mechanical movement of the neurological tissues as well as their sensitivity to mechanical stress or compression. These tests, along with relevant history and decreased range of motion, are considered by some to be the most important physical signs of disc herniation, regardless of the degree of disc injury. SLR is a neural tension test that can be used to rule in or out neural tissue involvement as a result of a space occupying lesion, often a lumbar disc herniation. It is one of the most common neurological tests of the lower limb
Oswestry Disability Index | 6th week
  Patient-completed questionnaire which gives a subjective percentage score of level of function (disability) in activities of daily living in those rehabilitating from low back pain. Most effective for persistent severe disability while the Roland-Morris is better for mild to moderate disability. Questionnaire examines perceived level of disability in 10 everyday activities of daily living

CONTACTS AND LOCATIONS:
Overall Officials: Nazish Rafique, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Max spine rehab centre, G8 markaz, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alexander CE, Weisbrod LJ, Varacallo MA. Lumbosacral Radiculopathy. 2024 Feb 27. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK430837/ PMID 28613587
- [Background] Berry JA, Elia C, Saini HS, Miulli DE. A Review of Lumbar Radiculopathy, Diagnosis, and Treatment. Cureus. 2019 Oct 17;11(10):e5934. doi: 10.7759/cureus.5934. PMID 31788391
- [Background] Chen BL, Guo JB, Zhang HW, Zhang YJ, Zhu Y, Zhang J, Hu HY, Zheng YL, Wang XQ. Surgical versus non-operative treatment for lumbar disc herniation: a systematic review and meta-analysis. Clin Rehabil. 2018 Feb;32(2):146-160. doi: 10.1177/0269215517719952. Epub 2017 Jul 17. PMID 28715939
- [Background] Shin JS, Lee J, Lee YJ, Kim MR, Ahn YJ, Park KB, Shin BC, Lee MS, Ha IH. Long-Term Course of Alternative and Integrative Therapy for Lumbar Disc Herniation and Risk Factors for Surgery: A Prospective Observational 5-Year Follow-Up Study. Spine (Phila Pa 1976). 2016 Aug 15;41(16):E955-E963. doi: 10.1097/BRS.0000000000001494. PMID 26882505
- [Background] Schoenfeld AJ, Laughlin M, Bader JO, Bono CM. Characterization of the incidence and risk factors for the development of lumbar radiculopathy. J Spinal Disord Tech. 2012 May;25(3):163-7. doi: 10.1097/BSD.0b013e3182146e55. PMID 22543563
- [Background] Abdurrahman G, Şener Ü, Karabacak H, Kağan Ü. Kadın ve erkek genç erişkinler arasında fiziksel aktivite ve yaşam kalitesi farklılıklarının araştırılması. Kocatepe Tıp Dergisi. 2011;12(3):145-50.
- [Background] Demirel A, Yorubulut M, Ergun N. Regression of lumbar disc herniation by physiotherapy. Does non-surgical spinal decompression therapy make a difference? Double-blind randomized controlled trial. J Back Musculoskelet Rehabil. 2017 Sep 22;30(5):1015-1022. doi: 10.3233/BMR-169581. PMID 28505956
- [Background] Oh H-J, Jeon C-B, Jeong M-G, Choi S-J. The effects of spinal decompression therapy on pain and disability in patients with chronic low back pain. The Journal of Korean Physical Therapy. 2017;29(6):299-302.